CLINICAL TRIAL: NCT01379248
Title: Effect of Thrombus Aspiration in Patients With Myocardial Infarction Presenting Late After Symptom Onset
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Steffen Desch, MD, Priv. - Doz. Dr. med., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEMI-Late-Presenter
Record Dates: First submitted 2011-06-20; First posted 2011-06-23 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

ARMS (2):
- thrombus aspiration (Experimental): Manual thrombus aspiration with dedicated catheter (Export, Medtronic Inc. Minneapolis, Minnesota, USA)
  Interventions: Device: manual thrombus aspiration (Export catheter, Medtronic Inc. Minneapolis, Minnesota, USA)
- no thrombus aspiration (No Intervention)

INTERVENTIONS:
Device: manual thrombus aspiration (Export catheter, Medtronic Inc. Minneapolis, Minnesota, USA) — manual thrombus aspiration catheter to be used during percutaneous coronary intervention
  Arms: thrombus aspiration

SUMMARY:
The purpose of this study is to examine the benefit of thrombus aspiration in patients with ST-elevation myocardial infarction presenting late after symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* ST-elevation myocardial infarction >12 and <48 hours after symptom onset
* age 18 to 90 years
* informed consent

Exclusion Criteria:

* prior fibrinolysis
* severe comorbidities with limited life expectancy
* pregnancy
* patient unable to give informed consent
* participation in another trial
* contraindications for heparin, aspirin or thienopyridines
* contraindications for cardiac magnetic resonance examination

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2011-06; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Microvascular obstruction (cardiac magnetic resonance imaging) | 1-4 days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leipzig Heart Center, Leipzig, Germany

REFERENCES:
- [Derived] Desch S, Stiermaier T, de Waha S, Lurz P, Gutberlet M, Sandri M, Mangner N, Boudriot E, Woinke M, Erbs S, Schuler G, Fuernau G, Eitel I, Thiele H. Thrombus Aspiration in Patients With ST-Segment Elevation Myocardial Infarction Presenting Late After Symptom Onset. JACC Cardiovasc Interv. 2016 Jan 25;9(2):113-22. doi: 10.1016/j.jcin.2015.09.010. PMID 26793952